Dose constraints for the temporal lobes during the optimization of intensity-modulated radiotherapy treatment plans for nasopharyngeal carcinoma

#### **Background**

Nasopharyngeal carcinoma (NPC) is common among Asians, especially in Southern China. Radiotherapy (RT) has been the mainstay of treatment for patients with non-disseminated NPC due to its anatomic location and radiosensitivity. In the management of the complex c

Intensity-modulated RT \MXT) is a major breakthrough in the treatment of NPC, and it was capable of producing \(\text{in}\) 's conformal dose distributions with steep dose gradients and complex isodose surfaces [31.7] he design of appropriate do e constraints for the organs at risk (OAR) during the optimization of IMRT treatment plane can enable significantly better OAR sparing and reduce subsequent complications. IMRT \(\text{in}\) inique can reduce the volume of high dose areas in the temporal lobes and thereby reduce risk of toxicities, compared with 2D-CRT [4, 5].

IMRT offers detailed to imetric parameters for temporal lobes based on dose-volume histogram (DVH). Some stules investigated the correlation between the incidence of TLI and IMRT dosimetric parameters. A retrospective study reported by Su et al. demonstrated that the 5-year incidence of TLI for a maximum dose of 64-68Gy or D1cc (the dose delivered to the 1 cubic centimeter volume, Gy) of 52-58 Gy was less than 5.0% after IMRT [6]. Similarly, a recent retrospective analysis of 20 patients with NPC and unilateral TLI showed that a dose of 69 Gy delivered to D0.5cc may be the dose tolerance of the temporal lobes after IMRT [7]. In our previous

study, we reported that the D1cc was the only independent predictor for radiation-induced TLI and estimated that the biologically equivalent tolerance doses at 2 Gy for the 5%,10% and 50% probabilities at 5 years to develop TLI were 62.83 Gy equivalents, 66.67Gy equivalents and 77.58 Gy equivalent, respectively [8]. However, only a few publications have quantified the risk of TLI complications in terms of normal tissue complication probability (NTCP) models.

Recently, we apply on five NTCP models, including (1) Lyman model and (2) logit-formula with dose-volume histogram (DVH) reduced to generalized equivalent uniform dose (EUD), (3) serial reconstruction unit (RU) model, (4) Poisson-EUD model, and (5) mean dose model for TLI to a population of 351 NPC patients treated with IMRT. As assessed qualitatively and quantitatively, the Lyman-EUD model fitted the data very well. The tolerance dose (TD) for the 5% and 10% probabilities of TLI development were 77 Gy and 80.4 Gy for Dm  $^{\circ}$ , in 2-Gy fractions ( $\alpha/\beta$  ratio, 3) in the current study (Manuscript has not been published).

According to the ICRU 83 report [9], overlap bety cervice planning target volume (PTV) and the planning organ at risk volume (PRV) leads to value that is shared by two contoured volumes. A conflict can occur if the planning aims of the verlapping contoured volume lack a common desired absorbed-dose range. To ensure the be onflict does not occur in a planning aims, at least two different methods can be applied. One method is based on subgivision of the volumes. Subdivision of the PTV of the gross targety plume (PTVnx) into region, with different prescribed absorbed doses (PTVsv1,PTVsv2, 17 /s /2 is the overlaps between PTVnx and temporal lobe) can be used in cases for which the PTVnx overlaps temporal 1 be. When the volume of PTVsv2 is less than 0.2 cubic centimeter (cc), the prescribe dose for FTV sv2 is as the same as that of the PTVsv1, D1cc 63.1Gy, Dmax 72.9Gy for TL (32 fractions) When the volume of PTVsv2 is between 0.2 cc and 0.5cc, the prescribe dose for PTVsv2 \( \) 66Gy, D1cc 63.1Gy, Dmax 72.9Gy for TL (32 fractions). When the volume of PTVsv2 is believeen 0.5 cc and 1cc, the prescribe dose for PTVsv2 is 66Gy, D1cc 65.8Gy, Dmax 75.2Gy for 31 (32 fractions). A study by Ng et al. showed that the 5-year local failure-free rate dropp a to 54% if more than 3cc volume within the gross primary tumor was under-dosed to below 6.5 Gy, compared with 90% in patients with smaller under-dosed volumes [10]. So, it is reasonable that prescribe dose for PTVsv2 is 66 Gy. The purpose of this prospective study is to evaluate the feasibility of dose constraints based on D1cc and Dmax for the temporal lobes following IMRT for NPC.

### Reference

- [1] Lee AW, Law SC, Ng SH, et al. Retrospective analysis of nasopharyngeal carcinoma treated during 1976–1985: late complications following megavoltage irradiation. Br J Radiol 1992;65:918-28.
- [2] Lee AW, Foo W, Chappell R, et al. Effect of time, destand fractionation on temporal lobe necrosis following radiotherapy for nasopharyngeal common. Int J Radiat Oncol Biol Phys 1998;40:35-42.
- [3] Xia P, Fu KK, Wong GW, et al. Cor crack on of treatment plans in obling intensity modulated radiotherapy for nasopharyngeal crack of a. Int J Radiat Oncol Pic Thys 2000,48(2):329-37.
- [4] Kam MK, Chau RM, Sue. J, Choi PH, Teo PM (2003), Litensity-modulated radiotherapy in nasopharyngeal carcinology in simetric advantage over conventional plans and feasibility of dose escalation. Int J Pacia, Chool Biol Phys 2003;56: 145-57.
- [5] Zhou GQ, Yu XL, Chen M, et al. Rachati in induced temporal lobe injury for nasopharyngeal carcinoma: a comparison of intensity in or ulated radiotherapy and conventional two-dimensional radiotherapy. Plos One 2013;8(7): 67 488.
- [6] Su SF, Huang Y, Xiao W W, et al. Clinical and dosimetric characteristics oftemporal lobe injury following intensity no ulated radiotherapy of nasopharyngeal carcinoma. Radiother Oncol 2012;104(3):312-3-5.
- [7] Sun Y, Zi ou GQ, Qi ZY, et al. Radiationinduced temporal lobe injury after intensity modulated radiocler py in nasopharyngeal carcinoma patients: a dose-volume-outcome analysis. BMC Cancer 2013;13:397.
- [8] Zeng L, Huang SM, Tian YM, et al. Normal Tissue Complication Probability Model for Radiation-induced Temporal Lobe Injury after Intensity-modulated Radiation Therapy for



Nasopharyngeal Carcinoma. Radiology 2015;276(1):243-9.

[9] Hodapp N. The ICRU Report 83: prescribing, recording and reporting photon-beam intensity-modulated radiation therapy (IMRT). Strahlenther Onkol 2012;188(1):97-99.

[10] Ng WT, Lee MC, Chang AT, et al. The impact of dosimetric inadequacy on treatment outcome of nasopharyngeal carcinoma with IMRT. Oral Oncol 2014;50:506512.

#### **Inclusion Criteria:**

- Newly-diagnosed and confirmed histopathologic diagnosis of nasopharyngeal squamous cell carcinoma, types WHO II-III, Stage I-IVA (AJCC staging 2017, 8th edition), treated with intensity-modulated radiotherapy.
- No head and neck surgery of the primary tv.nor rymph nodes except for incisional or excisional biopsies.
- Age between 18 years and 70 years
- Karnofsky score ≥80
- WBC 4,000/ul, platelet > 1c0,000/ul; serum creatinine < 1.6 mg/dl or 24hr. calculated creatinine clearance > 01.1/min.
- Must undergo pro treatment evaluation of tu nor extent and tumor measurement Tumor may be measurable or evaluable.
- Signed study-specific consent form proor to study entry.

# **Exclusion Criteria:**

- Stage IVB
- Evidence of all ant metastases
- Previous ir adiation for head and neck tumor  $\leq 6$  months prior to study entry
- Privious chemotherapy  $\leq 6$  months prior to study entry
- Patient is on other experimental therapeutic cancer treatment
- Other malignancy except non-melanoma skin cancer or a carcinoma not of head and neck origin and controlled at least 5 years



- Active untreated infection

- Major medical or psychiatric illness, which in the investigator's opinions, would interfere with

either the completion of therapy and follow-up or with full and complete understanding of the

risks and potential complications of the therapy

- Pregnant women

**Pretreatment evaluation** 

Each patient must have completed the following studies within six weeks prior to study entry

unless otherwise indicated.

Complete history and physical exam including weight and performance status.

Complete diagrammatic and descriptive documentation of the man ntof the primary and regional

(if any) following appropriate endoscopic procedures.

Complete dental and nutritional evaluation. Any provided dental repairs must be made and

prophylaxis instituted prior to radiotherapy.

Completion of the following laboratory st. Jies within 14 days of study mary: CBC and platelet

count; serum creatinine, creatinine reals ice, BUN, EBV-DNA, real pregnancy test for women.

Completion of the followin. Laboratory studies within six weeks of study entry: liver function

tests including AST, biling n. alkaline phosphatase.

Completion of the 11 owing radiologic studies within 6 weeks prior to study entry:

Chest CT scan

An MRI of head and neck with 71 vo trast with gadolinium and T2 sequences is required.

Abdominal ultrasonography

Bon scan

Radiotherapy

All patients were immobilized in the supine position with a thermoplastic mask. After

administration of intravenous contrast material, 3mm CT slices were acquired from the head to the

leve. 2cm below the sternoclavicular joint. Target volumes were delineated according to the

International Commission on Radiation Units and Measurements Reports(ICRU)50 and 62. The

primary nasopharyngeal gross tumor volume (GTVnx) and the involved cervical lymph nodes were

determined from the imaging, clinical, and endoscopic finding. The enlarged retropharyngeal nodes were outlined, together with primary GTV, as the (GTVnx) on the IMRT plans. The first clinical tumor volume (CTV1) was defined as the GTVnx plus a margin of 5-10mm for potential microscopic spread, including the entire nasopharynx mucosa plus a 5mm submucosal volume. The second CTV (CTV2) was defined by adding a margin of 5-10mm to CTV1 ( when CTV2 was adjacent to critical organs such as brain stem and spinal cord, the margin was reduced to 3-5mm) and included the retropharyngeal lymphnodal regions, clivus, skull base, pterygoid fossae, parapharyngeal space, inferior sphenoid sinus, and posterior edge of the nasal cavity and maxillary sinuses. The upper neck was also included in CTV2. Elective level IB irradiation was decided by the attending physician. The lower neck and the supraclavicular fossae were treated with a single anterior split field by conventional RT. Planning target volumes(F (")"s) for all gross tumor volumes and CTVs were generated automatically after delineation of tumor targets according to the immobilization and localization uncertainties. A sixtuan outsintegrated boost method was used. The prescribe dose was 66-70Gy to the PTV the Larvay FVnx, 60Gy to the PTV of CTV1(i.e., highrisk regions),54-56Gy to the PTV of CT 12 ..., low-risk regions),and G-70Gy to the PTV of the GTVnd for the metastatic cervical 1, 1, 21, lodes in 30-33 fraction. Let he GTV and CTV, the target volumes that received more than 55% of the prescribed dose was used to reflect the target coverage. The dose received by each an earl organ except temporal be was limited to tolerance according to the RTOG 0225 process

Dose constraints for the temporal lobes: Die; was the only independent predictor for radiation-induced TLI and estimated that the biologically equivalent tolerance doses at 2 Gy for the 5% and 10% probabilities at 5 years to de of p TLI were 62.83 Gy equivalents and 66.67Gy equivalents, respectively The tolerance dose (TD) for the 5% and 10% probabilities of TLI development were 77 Gy and 80.4 Gy for 2 max in 2-Gy fractions (α/β ratio, 3). These D1cc and Dmax of temporal lobes are convened to different dose constraints based on different fractions. Subdivision of the PTV of the cross target volume (PTVnx) into regions with different prescribed absorbed doses (PTV-10, 2TVsv2, PTVsv2 is the overlaps between PTVnx and temporal lobe) can be used in cases for which the PTVnx overlaps temporal lobe (Figure 1). For example, when the volume of PTVsv2 is less than 0.2 cubic centimeter (cc), the prescribe dose for PTVsv2 is as the same as that of the PTVsv1, D1cc 62.0Gy, Dmax 71.5Gy for TL (30 fractions), D1cc 63.1Gy, Dmax 72.9Gy for TL (32

fractions) and D1cc 63.7Gy, Dmax 73.6Gy for TL (33 fractions), respectively. When the volume of PTVsv2 is between 0.2 cc and 0.5cc, the prescribe dose for PTVsv2 is 66Gy, D1cc 63.1Gy, Dmax 72.9Gy for TL (32 fractions), D1cc 63.7Gy, Dmax 73.6Gy for TL (33 fractions), respectively. When the volume of PTVsv2 is between 0.5 cc and 1cc, the prescribe dose for PTVsv2 is 66Gy, D1cc 65.8Gy, Dmax 75.2Gy for TL (32 fractions), D1cc 66.4Gy, Dmax 75.9Gy for TL (33 fractions), respectively (Table 1). If the volume of PTVsv2 is more than 1cc, dose constraints for temporal lobes is not protocolized, and is based on the discretion of the attending physician in individual cases.



Figure 1 Subdivision of the PTV of the gross target volume (PTVnx) into regions with different prescribed absorbed doses (PTVsv1,PTVsv2, PTVsv2 is the overlaps between PTVnx and temporal lobe) can be used in cases for which the PTVnx overlaps temporal lobe.

Table 1. The relationship between dose constraints for the temporal lobes and the incidence of temporal lobe injury (TLI).

| Total dose70Gy/fractions | Incidence of TLI | Volume of TL D1cc | TL Dmax |
|--------------------------|------------------|-------------------|---------|
| 30 | 5% | 62.0 | 71.5 |
| | 10% | 61.5 | 73.7 |
| 32 | 5% | 53.1 | 72.9 |
| | 10% | 65.8 | 75.2 |
| 33 | 5% | 63.7 | 73.6 |
| | 10.0 | 66.4 | 75.9 |

# Chemotherapy

Chemotherapy included or new cut chemotherapy, concurrent chemotherapy combined with induction chemotherapy a valor adjuvant chemotherapy. The regimens of induction chemotherapy and adjuvant chemotherapy included docetaxel and cisplatin (DP), gemcitabine and cisplatin (GP) and 5-Fu and cisplatin (PF). The DP protocol consisted of docetaxel 75mg/m2 IV on day 1, cisplatin 75 mg/m2 on day1. The GP protocol consisted of gemcitabine 1.0g/m2 IV on day 1, 8, cisplatin 75 mg/m2 on day1. The PF protocol consisted of cisplatin 80mg/m2 IV on day 1 and 5-Fu 800mg/m2d continuously IV on day 1-5. For patients who receive induction chemotherapy, both DP, GP and PF are repeated every 3 weeks for 2-3 cycles. This is followed by cisplatin 30mg/m2 IV weekly or

cisplatin 80mg/m2 IV on day1,22 during radiation. For patients who received adjuvant chemotherapy, regimens are repeated every 3 week for 3cycles. Chemotherapy is not protocolized and is used at the discretion of the attending physician in individual cases.

# Follow up

After the completion of radiotherapy, all patients will be followed up every 1-3months during the first 2 years, every 6 months in years 2 to 5 and annually thereafter. During the follow-up sessions, disease status and treatment toxicity will be assessed by performing MRI to the head and neck region, chest radiograph, abdominal ultrasonograph, and physical examination. When indicated, as well as whole-body bone scan if required.

### Statistical analysis

The sample size will be adjusted by 20% to account or patients that die within the 5 years and are not evaluable for the toxicity endpoint, at a for ineligible or inevaluable to data) cases. The total target accrual is 350 patients. The survey of time is measured from Data of RT completion to the date of the event or last follow up visit. All analyses will be a proportional with SPSS software, version 19.0. The Kaplan-Me. or method is used to calculate the overall survival (OS), local recurrence-free survival (ACS) rates. Multivariate unalysis will be done by using the Cox proportional hazard more independent are nectors among various side effects.

